CLINICAL TRIAL: NCT05040048
Title: Taxonomy of Neurodegenerative Diseases : Observational Study in Alzheimer's Disease and Parkinson's Disease (AETIONOMY)
Brief Title: Taxonomy of Neurodegenerative Diseases : Observational Study in Alzheimer's Disease and Parkinson's Disease
Acronym: AETIONOMY
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Innovative Medicines Initiative (Other); Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other); ICM Co. Ltd. (Industry); University Hospital, Bonn (Other); Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: 14-37; 2015-A00356-43 (Registry Identifier: ID RCB)
Record Dates: First submitted 2015-07-24; First posted 2021-09-10 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Alzheimer's Disease; Parkinson's Disease
Keywords: Alzheimer; Parkinson; Data mining; Biomarkers; Stratification
MeSH Terms: conditions — Alzheimer Disease; Parkinson Disease | interventions — Biological Products

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood and CSF samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Parkinson's disease Group: Blood, cerebrospinal fluid (CSF) and skin biopsy samples. Neuropsychological assessment. Motor and non motor assessments for Parkinson's disease group only.
  Interventions: Other: Clinical, biological and imaging assessment
- Alzheimer's disease Group: Blood, cerebrospinal fluid (CSF) and skin biopsy samples. Neuropsychological assessment. Brain MRI for Alzheimer's disease group only.
  Interventions: Other: Clinical, biological and imaging assessment

INTERVENTIONS:
Other: Clinical, biological and imaging assessment

SUMMARY:
The AETIONOMY project will generate a refined taxonomy and testable mechanisms underlying the derived stratification of patients.

DETAILED DESCRIPTION:
The main objective of the AETIONOMY clinical study is to test in real clinical samples the validity of the hypothesized underlying pathogenic mechanisms of AD and PD.

Although not fully understood, the pathophysiology of neurodegenerative diseases results from the complex interplay between several biological pathways such as neuronal excitotoxicity, oxidative stress, protein miss-folding and aggregation, neuroinflammation, apoptosis etc. It is thus likely that the maps generated by the AETIONOMY project will comprise several distinct biological hypotheses and subgroups of patients defined by 1 or more of these hypotheses. The Consortium has insufficient resources to validate all these hypotheses. Although it is anticipated that the AETIONOMY Project will provide novelty in the investigators' understanding of neurodegenerative diseases, it is expected that previously known biological pathways will come out from the data mining approach, e.g. mitochondrial pathway for PD or beta-amyloid aggregation for AD. AETIONOMY project will take advantage of these previously known pathways that will be considered as internal controls. One or two novel pathogenic pathways will be tested in parallel. Overall, this strategy will allow validating two hypotheses for each neurodegenerative disease (AD and PD). As it cannot be predicted what hypotheses will precisely rise from the data mining, the approach must be adaptative. However, it is possible to anticipate which population, clinical data, brain imaging procedure, and which biological samples will have to be applied for their validation. The AETIONOMY clinical study thus aims at assembling a standardized clinical, brain imaging, and biological collection from AD patients, PD patients and healthy controls to validate the model proposed by the AETIONOMY project. The Consortium will identify potential pathogenic pathways (established and novel) involved in AD and PD and will deliver surrogate markers which serve as readouts of the involved pathways. The model will be considered validated if the selected makers allow subject stratification in the AETIONOMY clinical study according to what has been postulated in the model. Additional correlation between biomarker expression and brain imaging will be performed when available. A transversal cohort will be recruited from 4 sites in Europe (France, Germany, Spain, and Sweden), including AD and PD patients, individuals at risk of AD and PD, and healthy controls.

Approximately 655 subjects will be recruited. Subjects will have a single study visit with clinical assessments, biological sampling, brain imaging (AD group only). Standardized procedures will be used for biological sampling as well as for brain image acquisition.

ELIGIBILITY:
INCLUSION CRITERIA

FOR ALL

* Male or female.
* Ability to provide written informed consent in accordance with International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH), Good Clinical Practice (GCP) and local regulations.
* Have social security insurance (for French patients only).

PARKINSON'S DISEASE GROUP

Idiopathic PD patients:

* 40 ≤ Age ≤75 years.
* Diagnosed as "clinically possible", "clinically probable" or "clinically definite" idiopathic PD according to UK Parkinson's Disease Society Brain Bank (UKPDSBB, Hugues et al. 1992).
* A diagnosis of PD for strictly 5 years or less at inclusion.

PD patients with mutation in Parkin, Leucine-rich repeat kinase 2 (LRRK2) or Glucosidase beta acid (GBA) gene:

* Age ≥ 18 years.
* Diagnosed with PD and genotyped for a mutation in Parkin, LRRK2 or GBA genes.

Subjects at risk of PD:

* Age ≥ 18 years.
* No clinical symptom of PD at neurological examination (akinesia, no extrapyramidal rigidity, and no rest tremor).
* One of the following criteria: First-degree relative of a PD index case with a LRRK2 or GBA mutation OR Idiopathic Rapid eye movement (REM) Behavior Disorder (RBD) as defined by the presence of at least 1 of the following conditions: (1) Potentially harmful dream-enacting behaviors in response to dream content and loss of normal electromyographic (EMG) atonia on polysomnography (PSG) manifest as sustained muscle activity during more that 27% of REM sleep in the chin EMG; (2) Abnormal behavior during REM sleep .

Healthy control subjects:

* Age ≥ 18 years.
* Normal neurological examination.
* Absence of cognitive impairment defined as: Mini Mental State Examination (MMSE) score ≥ 26 and Objective cognitive performance within the normal range (performance within 1.5 SD) in all tests from a specific test battery.

ALZHEIMER'S DISEASE GROUP

Prodromal AD patients:

* Age ≥ 50 to ≤ 80 years.
* Study partner/caretaker has noticed a recent gradual decrease in the subject's memory (e.g. over the prior 12 months), which the subject may or may not be aware of.
* Cognitive requirements:

  * Abnormal memory function at screening based on the Free and Cued Selective Reminding Test (FCSRT-IR) of free recall <17 or total recall <40
  * Screening MMSE score of 26 or above
  * Screening global Clinical Dementia rating (CDR) of 0.5 with a memory box score of 0.5 or 1
  * Aside from memory impairment, general cognition and functional performance are largely preserved such that a diagnosis of AD with dementia cannot currently be made.
* CSF Aβ1-42 level ≤ 550 pg/mL as measured by the local laboratory (cut off may depend on the performing lab).
* Subject or study partner has ability to provide written informed consent in accordance with ICH, GCP, and local regulations.
* Each subject must have a study partner/caretaker who is reliable and competent. The study partner/caretaker must have a close relationship with the subject, have face to face contact at least 3 days/wk for a minimum of 6 waking hours/wk and be willing to accompany the subject to the study assessments.
* Be able to read at a 6th grade level or equivalent, as determined by the investigator, and must have a history of academic achievement and/or employment sufficient to exclude mental retardation.
* Have results of clinical laboratory tests (complete blood count [CBC], blood chemistries, thyroid stimulating hormone [TSH]) within normal limits or clinically acceptable to the site principal investigator at screening.
* Have results of a physical examination, vital signs, and electrocardiogram (ECG) within normal limits or clinically acceptable to the site principal investigator at screening.

Preclinical AD patients (asymptomatic at risk of AD):

* Age ≥ 50 to ≤ 80 years.
* Subjects with no cognitive impairment: MMSE scores ≥ 26 and Objective cognitive performance within the normal range (performance within 1.5 SD) in all tests from a specific test battery and CDR scale score of 0
* CSF Aβ1-42 level ≤ 550 pg/mL as measured by the local laboratory (cut off may depend on the performing lab).
* Ability to provide written informed consent in accordance with ICH, GCP, and local regulations

Healthy control subjects:

* Age ≥ 50 to ≤ 80 years.
* Normal neurological examination.
* Absence of cognitive impairment, defined as: MMSE score ≥ 26 and Objective cognitive performance within the normal range (performance within 1.5 SD) in all tests from a specific test battery and CDR scale score of 0
* CSF Aβ1-42 level ≥ 550 pg/mL as measured by the local laboratory (cut off may depend on the performing lab).
* Ability to provide written informed consent in accordance with ICH, GCP, and local regulations.

EXCLUSION CRITERIA

FOR ALL

* Any of the following medications within 1 week prior to inclusion:

  * Anti-inflammatory
  * Anti-neoplastic
  * Immunosuppressives
  * Systemic corticosteroids
* Vaccination with live vaccines within 3 weeks and/or with inactivated vaccines within 2 weeks prior to inclusion
* On-going viral or bacterial infection requiring at least symptomatic treatment, or antibiotics, or associated with fever or pain.
* Any psychiatric condition, which in the opinion of the investigator might preclude participation.
* Any lab abnormality, which in the opinion of the investigator might preclude participation.
* Pregnant woman or lactating or planning pregnancy during the course of the study (Includes a negative urine pregnancy test or to be of non-child bearing potential).
* Participant who does not wish to be informed of any clinically relevant abnormalities (as determined by the investigator at that site) identified during the course of the study (For France only).

PARKINSON'S DISEASE GROUP

Idiopathic PD patients:

* Family history of PD.
* Atypical PD syndromes due to either drugs (e.g., metoclopramide, flunarizine, neuroleptics) or metabolic disorders (e.g., Wilson's disease), encephalitis, or degenerative diseases (e.g., progressive supranuclear palsy).
* Currently taking neuroleptics or has taken neuroleptics within 6 months of baseline.
* Under guardianship or curatorship.

PD patients with mutation in Parkin, LRRK2 or GBA gene:

* Atypical PD syndromes due to either drugs (e.g., metoclopramide, flunarizine, neuroleptics) or metabolic disorders (e.g., Wilson's disease), encephalitis, or degenerative diseases (e.g., progressive supranuclear palsy).
* Currently taking neuroleptics or has taken neuroleptics within 6 months of baseline.
* Under guardianship or curatorship.

Subjects at risk of PD:

* Clinically significant abnormal neurological examination (in the opinion of the investigator).
* A clinical diagnosis of PD as determined by the investigator.
* Currently taking neuroleptics or has taken neuroleptics within 6 months of baseline.
* Under guardianship or curatorship.

PD Healthy control subjects:

* A recent or ongoing, uncontrolled, clinically significant medical condition within 3 months of screening (such as, but not limited to, diabetes, hypertension, thyroid or endocrine disease congestive heart failure, angina, cardiac or gastrointestinal disease)
* Current or active clinically significant neurological disorder (in the opinion of the investigator).
* First-degree relative with idiopathic PD (parent, sibling, child).
* Received any drugs that might interfere in the opinion of the investigator with neurological and cognitive assessments: for example neuroleptics, benzodiazepine or antidepressant.
* Under guardianship or curatorship.

ALZHEIMER'S DISEASE GROUP

Prodromal AD patients:

* Rosen-modified Hachinski Ischemia Score > 4 at screening (ie, evidence of vascular dementia).
* Known history of stroke or evidence from MRI scan that is clinically important in the investigator's opinion.
* Evidence of a clinically relevant neurological disorder other than the disease being studied (ie, probable AD), including but not limited to: vascular dementia, parkinsonism, frontotemporal dementia, Huntington's disease, amyotrophic lateral sclerosis, multiple sclerosis, progressive supranuclear palsy, neurosyphilis, dementia with Lewy bodies, other types of dementia, mental retardation, hypoxic cerebral damage, cognitive impairment due to other disorders, or head trauma with loss of consciousness that led to persistent cognitive deficits.
* The subject has evidence of a clinically relevant or unstable psychiatric disorder, based on Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition - Text Revision (DSM-IV-TR) criteria,
* Previous MRI scan showing evidence of a neurological disorder other than probable AD or > 4 cerebral microhemorrhages (regardless of their anatomical location or diagnostic characterization as "possible" or "definite"), a single area of superficial siderosis, evidence of a prior macrohemorrhage, 3 lacunar infarcts, any cortical infarct over 5 mm, or any other clinically significant finding (eg, brain tumor).
* A recent or ongoing, uncontrolled, clinically significant medical condition within 3 months of the screening (such as, but not limited to, diabetes, hypertension, thyroid or endocrine disease congestive heart failure, angina, cardiac or gastrointestinal disease)
* The subject has:

  1. a history of clinically significant vitamin B12 or folate deficiency in the 6 months immediately before Screening, or
  2. vitamin B12 or folate deficiency in addition to increased serum homocysteine or methylmalonic acid levels at screening.
* Contraindications for MRI scan (pacemaker, implanted cardioverter-defibrillator, neurostimulation system, cochlear implant, metallic foreign body (metal sliver) in the eye, metallic prosthesis, cerebral aneurysm clip, ventriculoperitoneal neurosurgical bypass valve, fixed dental prosthesis, known claustrophobia).
* Contraindications for lumbar puncture: current treatment with anticoagulants (e.g., coumadin, heparin) or double antiaggregant therapy.

Preclinical AD patients (asymptomatic at risk of AD):

* Rosen-modified Hachinski Ischemia Score > 4 at screening (ie, evidence of vascular dementia).
* Known history of stroke or evidence from MRI scan that is clinically important in the investigator's opinion.
* Evidence of a clinically relevant neurological disorder other than the disease being studied (ie, probable AD), including but not limited to: vascular dementia, parkinsonism, frontotemporal dementia, Huntington's disease, amyotrophic lateral sclerosis, multiple sclerosis, progressive supranuclear palsy, neurosyphilis, dementia with Lewy bodies, other types of dementia, mental retardation, hypoxic cerebral damage, cognitive impairment due to other disorders, or head trauma with loss of consciousness that led to persistent cognitive deficits.
* The subject has evidence of a clinically relevant or unstable psychiatric disorder, based on DSM-IV-TR criteria,
* Previous MRI scan showing evidence of a neurological disorder other than probable AD or > 4 cerebral microhemorrhages (regardless of their anatomical location or diagnostic characterization as "possible" or "definite"), a single area of superficial siderosis, evidence of a prior macrohemorrhage, 3 lacunar infarcts, any cortical infarct over 5 mm, or any other clinically significant finding (eg, brain tumor).
* The subject has:

  1. a history of clinically significant vitamin B12 or folate deficiency in the 6 months immediately before Screening, or
  2. vitamin B12 or folate deficiency in addition to increased serum homocysteine or methylmalonic acid levels at screening.
* Contraindications for MRI scan (pacemaker, implanted cardioverter-defibrillator, neurostimulation system, cochlear implant, metallic foreign body (metal sliver) in the eye, metallic prosthesis, cerebral aneurysm clip, ventriculoperitoneal neurosurgical bypass valve, fixed dental prosthesis, known claustrophobia).
* Contraindications for lumbar puncture: current treatment with anticoagulants (e.g., coumadin, heparin) or double antiaggregant therapy.
* Under guardianship or curatorship.

AD Healthy control subjects:

* A recent or ongoing, uncontrolled, clinically significant medical condition within 3 months of screening (such as, but not limited to, diabetes, hypertension, thyroid or endocrine disease congestive heart failure, angina, cardiac or gastrointestinal disease)
* Current or active clinically significant neurological disorder (in the opinion of the investigator).
* Received any drugs that might interfere in the opinion of the investigator with neurological and cognitive assessments: for example neuroleptics, benzodiazepine or antidepressant.
* Contraindications for MRI scan (pacemaker, implanted cardioverter-defibrillator, neurostimulation system, cochlear implant, metallic foreign body (metal sliver) in the eye, metallic prosthesis, cerebral aneurysm clip, ventriculoperitoneal neurosurgical bypass valve, fixed dental prosthesis, known claustrophobia).
* Contraindications for lumbar puncture: current treatment with anticoagulants (e.g., coumadin, heparin) or double antiaggregant therapy, clinically significant coagulopathy or thrombocytopenia.
* Under guardianship or curatorship.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: PD GROUP (n=325):
  * 240 idiopathic PD patients
  * 40 PD patients with mutations of the gene of Parkin (n =10), LRRK2 (n=10) and GBA (n=20)
  * 45 subjects at risk of PD:
    * first degree relative of a PD index case with mutation (LRRK2, n=10)
    * first degree relative of a PD index case with risk factor (GBA, n=10)
    * subjects with idiopathic RBD (n=25)
  AD GROUP (n=150):
  * 90 prodromal AD patients
  * 60 preclinical AD patients
  HEALTHY CONTROLS (n=180):
  * 90 healthy controls matched for age and sex for PD group's subject
  * 90 healthy controls matched for age and sex for AD group's subject
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2015-09-04 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Performance of the biomarker in discriminating between the taxonomy of interest and the remainder of the AD/PD subjects | 27 months
  assessments of the effectiveness of a biomarker in assigning a taxonomy will be made using subjects with the taxonomy membership of interest and the Healthy Controls. biomarkers), surrogate of a causative mechanism for PD or AD (2 biomarkers for each disease).
  AETIONOMY is built to validate the mechanism-based stratification of patients by testing in real clinical samples the hypotheses underlying pathogenic mechanisms identified by the consortium. It is expected to assess a large panel of biomarkers exploring biocollections (blood, DNA, CSF, skin biopsies) and imaging, associated with clinical assessment: (Pathway-Material for assessment (planned biomarker)) Astroglial inflammation-CSF(YKL40) Neuroinflammation-CSF and/or blood(MRP8, MRP14) Cross-talk mitochondria/neuroinflammation-CSF(TFAM, HSD10) Epigenetics-DNA(SNCA methylation) Insulin pathway-CSF and/or blood(IRS) Stress-induced comorbidity-DNA(CRH, CRHR1, MAPT) Uptake of aggregate proteins-material TBD(Syndecan)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe CORVOL, MD, PhD, Principal Investigator — jean-christophe.corvol@aphp.fr
Locations (4):
- CIC Neurosciences - ICM - Hôpital Pitié-Salpêtrière, 47-83 Bd de l'Hôpital, Paris, France
- Universitaetsklinikum Bonn (UKB), Sigmund-Freud 25 Strasse, Bonn, Germany
- Institut d'Investigacions Biomediques August Pi i Sunyer (IDIBAPS), Rossello 149- 153, Barcelona, Spain
- Karolinska Institutet (KI), Karolinska University Hospital S3:01, Stockholm, Sweden